CLINICAL TRIAL: NCT07021716
Title: COVID-19 Knowledge, Attitudes, Practices and Perceived Risk: Cross Sectional Mixed Methods
Acronym: Coronavirus
Status: Completed | Type: Observational
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Aliza Bitton Ben-Zacharia, Assistant Professor, Hunter College of City University of New York
Other Study IDs: 24-08027786
Record Dates: First submitted 2025-06-09; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2020-12

CONDITIONS: COVID - 19; Multiple Sclerosis
Keywords: COVID; Knowledge; Attitudes; Practices
MeSH Terms: conditions — COVID-19; Multiple Sclerosis; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with multiple sclerosis: Patients with multiple sclerosis answered the KAP survey providing answers to open ended questions analyzed qualitatively.
  Interventions: Other: No Interventions
- Healthcare professionals: Healthcare professionals answered the KAP survey providing answers to open ended questions analyzed qualitatively.
  Interventions: Other: No Interventions
- Laypeople: Laypeople answered the KAP survey providing answers to open ended questions analyzed qualitatively.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No Interventions

SUMMARY:
Knowledge, attitudes, behaviors and perceived risk highlight the importance of education translated into actions to reduce the risk of global infections. The purpose was to investigate the knowledge, attitudes and practices (KAP), and perceived risk associated with COVID-19 among patients with multiple sclerosis (MS), healthcare providers and laypeople during the first 6-months of the pandemic. A descriptive, cross-sectional, partially mixed-methods explanatory sequential design was employed, using convenience sampling. Data were collected through a demographic and a KAP questionnaires including perceived risk assessment. Quantitative data were analyzed with descriptive and inferential statistics, while qualitative comments underwent thematic analysis.

DETAILED DESCRIPTION:
This is a descriptive cross-sectional, partially mixed method explanatory sequential study, following the Good Reporting of A Mixed Methods Study (GRAMMS) guideline. This study concentrated on the KAP of patients with MS, healthcare professionals and lay people. The aim was to explain the quantitative survey results with qualitative themes in an explanatory sequential design. The goal of the quantitative phase was to examine the COVID-19-related knowledge, attitudes, and practices among healthcare professionals, laypeople, and patients with multiple sclerosis (MS) during the first 6 months of the pandemic and to compare the perceived risk of coronavirus infection across these three groups. The goal of the qualitative phase of this study was to identify and analyze the emergent themes reflecting participants' perceptions of their risk related to COVID-19. The goal of the mixed methods phase was to generate integrated support for the participants knowledge, attitudes, practices, and perceived risk based upon quantitative and qualitative evidence.

Theoretical Framework. The knowledge-attitude-behavior (KAB) model considers that knowledge and information gained are fundamental prerequisite for behavioral changes. People are able to gain knowledge and practical skills through education. Accordingly, professionals, laypeople, and patients need to learn and get basic and advanced knowledge, which can lead to the growth of positive beliefs and attitudes that are fortified with the acceptance of healthy behaviors (Liu et al., 2016; Zulkifli et al., 2022). Furthermore, the KAB framework highlights the relationship between knowledge, attitudes and behaviors and their influence on actions (Maleki et al., 2020).

Instruments. The KAP questionnaire consisted of a demographic form, and a KAP questionnaire. The prequestionnaire solicited basic demographic information such as the participant's age, gender, education level, and patients' disease related information. The KAP instrument was adapted from the CDC (CDC; CDC Center for Disease Control; Maike WintersComments to Author 2017) and used with permission. The KAP survey instrument has been used nationally and internationally to explore people's health behaviors and their lifestyle changes (Azlan et al., 2020; CDC; Masoud et al., 2021; Qalati et al., 2023; Zhong et al., 2020). The survey included 50 close-ended questions that took 20-25 minutes to complete. It covered demographics (10 items), COVID-19 knowledge (15 items), attitudes (17 items), and practices (8 items). True/false questions had "I don't know" and "declined to answer" options, with responses categorized as correct or incorrect (Seninde & Chambers, 2021; Smyth et al., 2006). Open-ended questions were analyzed to assess the participants' perceptions qualitatively.

Perceived risk for contracting COVID-19 was assessed using a 5-point scale (0=no risk at all, 1=a small risk, 2=a moderate risk, 3=a high risk, 4=Don't know). Perceived risk of COVID was assessed as a categorical variable. It was analyzed as dichotomous variable (low risk vs. moderate/high risk) and as 4-categorical variable (low risk, moderate risk, high risk and don't know). Perceived risk was assessed and analyzed in each group, patients with MS, healthcare professionals and lay people.

Data Collection. The population for this study included healthcare professionals (nurses and physicians), patients with MS, and lay people from the northeast region in the USA. It included participants from New York, Connecticut and Massachusetts. A convenience sampling approach was used to enhance recruitment. The participants were recruited via blast emails through health centers, MS centers, and community resources. Data were collected via an online self-reported questionnaire from April 2020 to September 2020. The surveys were completed online via anonymous and confidential software, i.e., a 'Monkey' survey. The inclusion criteria of the study included adult people (≥18 years), consisting of patients with MS, healthcare professionals (nurses and physicians), and adult lay people. The project did not include any exclusion criteria.

Data Analysis. Descriptive analyses were used to characterize the sample. Chi-square and Kruskal Wallis tests assessed associations between demographics, KAPs, and perceived risk. Kruskal Wallis test compared KAP across patients with MS, healthcare professionals, and laypeople. Logistic regression assessed the perceived risk as a dependent dichotomized variable (low and moderate/high risk), immunocompromised state or vaccination hesitancy as independent variables controlling for age, sex, and education. Statistical significance was set at p<.05. A qualitative thematic analysis was performed and coded on participants' comments by two researchers (AB and JS) to identify key themes reaching data saturation.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of the study included adult people (≥18 years), consisting of patients with MS, healthcare professionals (nurses and physicians), and adult lay people.

Exclusion Criteria:

* The project did not include any exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population for this study included healthcare professionals (nurses and physicians), patients with MS, and lay people from the northeast region in the USA. It included participants from New York, Connecticut and Massachusetts. A convenience sampling approach was used to enhance recruitment. The participants were recruited via blast emails through health centers, MS centers, and community resources. Data were collected via an online self-reported questionnaire from April 2020 to September 2020. The surveys were completed online via anonymous and confidential software, i.e., a 'Monkey' survey. The inclusion criteria of the study included adult people (≥18 years), consisting of patients with MS, healthcare professionals (nurses and physicians), and adult lay people. The project did not include any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Knowledge | 6 months
  Knowledge associated with COVID-19
Perceived Risk | 6 months
  Perceived risk for contracting COVID-19 was assessed using a 5-point scale (0=no risk at all, 1=a small risk, 2=a moderate risk, 3=a high risk, 4=Don't know). Perceived risk of COVID was assessed as a categorical variable. It was analyzed as dichotomous variable (low risk vs. moderate/high risk) and as 4-categorical variable (low risk, moderate risk, high risk and don't know). Perceived risk was assessed and analyzed in each group, patients with MS, healthcare professionals and lay people.
Attitudes | 6 months
  Attitudes associated with COVID-19
Practices | 6 months
  Practices associated with COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter College, New York, New York, United States